CLINICAL TRIAL: NCT05693688
Title: Atosiban Versus Placebo in the Treatment of Late Threatened Preterm Birth
Brief Title: Atosiban Versus Placebo in the Treatment of Late Threatened Pre-term Birth
Acronym: APOSTEL 8
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Nottingham University Hospitals NHS Trust (Other); Amphia Hospital (Other); St. Antonius Hospital (Other); Deventer Ziekenhuis (Other); Erasmus Medical Center (Other); Flevoziekenhuis (Other); Franciscus Gasthuis (Other); Gelre Hospitals (Other); Groene Hart Ziekenhuis (Other); Isala (Other); Leiden University Medical Center (Other); Martini Hospital Groningen (Other); Maxima Medical Center (Other); Frisius Medisch Centrum (Other); Haaglanden Medical Centre (Other); Maastricht University Medical Center (Other); Medisch Spectrum Twente (Other); OLVG (Network); Radboud University Medical Center (Other); Rijnstate Hospital (Other); Spaarne Gasthuis (Other); Tergooi Hospital (Other); University Medical Center Groningen (Other); UMC Utrecht (Other); Diakonessenhuis, Utrecht (Other); Ziekenhuisgroep Twente (Other); Zuyderland Medical Centre (Other); National Maternity Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Martijn A. Oudijk, MD, PhD, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL80-84800-98-41027
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Preterm Birth
Keywords: preterm birth; threatened preterm birth; preterm labour; atosiban; adverse neonatal outcome
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — atosiban

STUDY DESIGN:
Intervention Model Description: International, multicenter, double blinded, placebo controlled RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- atosiban (Experimental): Atosiban: bolus injection of 6.75 mg/0.9 ml atosiban in one minute followed by a continuous infusion of 18 mg/hour (=24ml/hour) for 3 hours followed by a continuous infusion of 6 mg/hour (=8 ml/hour) for the remaining 45 hours.
  Interventions: Drug: Atosiban
- placebo (Placebo Comparator): Placebo: injection of 0.9 ml saline in one minute followed by a saline infusion for 3 hours (24 ml/hour) followed by a continuous infusion (8 ml/hour) for the remaining 45 hours.
  Interventions: Drug: Atosiban

INTERVENTIONS:
Drug: Atosiban — atosiban i.v. administred for 48 hours. The medication will be administered by a bolus injection of 6.75 mg/0.9 mL in 1 min followed by a continuous infusion of 18 mg/hour for 3 hours followed by a continuous infusion of 6 mg/hour for the remaining 45 hours.
  Other Names: Tractocile

SUMMARY:
The aim of this study is to investigate if tocolysis with atosiban in late preterm birth (30 to 34 weeks) is (cost-) effective compared with placebo in improving neonatal morbidity and mortality.

DETAILED DESCRIPTION:
Research question Does tocolysis with atosiban reduce neonatal mortality and mortality in women with threatened preterm birth between 30 and 34 weeks when compared to placebo?

Study design Multicenter, double blinded, placebo controlled RCT

Study population Women with threatened preterm birth between 30 and 34 weeks of gestation are eligible for the trial. More than 20 hospitals (including all 10 perinatal centres) in the Netherlands will participate in this trial, as well as 15 hospitals in the UK and 1 in Dublin, Ireland.

Threatened preterm birth is defined as listed below in the inclusion criteria. Our previous APOSTEL III study showed that half of the women with these criteria deliver within seven days, validating this definition of women at high risk for preterm birth.

Inclusion criteria

* Women ≥ 18 years old
* Singleton or twin pregnancy
* Gestational age between 30 0/7 and 33 6/7 weeks
* Threatened preterm birth defined by regular uterine contractions, AND one of the following:

  * Cervical length of < 15 mm OR
  * Cervical length of 15-30 mm and a positive Fibronectine test (≥ 50 ng/mL) OR
  * In case of absence of cervical length measurement in local protocol a positive Fibronectin test or Partus test OR
  * Ruptured amniotic membranes

Exclusion criteria

* Previous treatment for threatened preterm birth with corticosteroids.
* Contra-indication for tocolysis
* Signs of fetal distress
* Signs of intra uterine infection

Participants RCT: 760 (380 per group)

Description of intervention(s) Tocolysis with atosiban versus placebo.

Outcome measures The primary outcome is a combined perinatal outcome of severe neonatal morbidity and perinatal mortality Secondary outcomes will be birth within 48 hours, time to delivery, gestational age at delivery, birth weight, number of days on invasive mechanical ventilation, length of admission in NICU, convulsions, asphyxia, meningitis, pneumothorax and mortality until 3 months corrected age, maternal infection, maternal side effects and costs.

All outcomes are in the electronic patient file. No additional tests are required for mother or baby.

Power / data analysis Based on the APOSTEL 3 data, the proportion of adverse perinatal outcome in women randomized between 30 and 34 weeks gestation and treated with atosiban was 6%. Based on two recent studies, we expect a 49,8% reduction of 11,95% adverse perinatal outcome in the placebo group to 6% in the atosiban group. Therefore we need to randomize 722 women (beta-error 0.2; alpha error 0.05). Assuming a 5% drop-out rate, we need to randomize 760 women (380 in each arm).

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years
* Singleton or twin pregnancy
* Gestational age between 30 0/7 and 33 6/7 weeks
* Threatened preterm birth defined by regular uterine contractions, AND one of the following:

  * Cervical length of < 15 mm OR
  * Cervical length of 15-30 mm and a positive Fibronectine test (≥ 50 ng/mL) OR
  * In case of absence of cervical length measurement in local protocol a positive Fibronectin test or Partus test OR
  * Ruptured amniotic membranes

Exclusion Criteria:

* Previous treatment for threatened preterm birth with corticosteroids in current pregnancy
* Contra indication for tocolysis
* Signs of fetal distress
* Signs of intra uterine infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 760 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Adverse neonatal outcome | Up to 3 months corrected age
  Combination perinatal mortality and severe neonatal morbidity (BPD, NEC, ROP, IVH, PVL, sepsis,

SECONDARY OUTCOMES:
Birth within 48 hours | 48 hours
Time to delivery | Not applicible
Gestational age at delivery | At birth
Birth weight | At birth
Mechanical ventilation | Up to 3 months corrected age
  Number of days on invasive ventilation
NICU | Up to 3 months corrected age
  Lengt of admission in NICU
Convulsions | Up to 3 months corrected age
Asphyxia | Up to 3 months corrected age
Meningitis | Up to 3 months corrected age
Pneumothorax | Up to 3 months corrected age
Maternal infection | Up to 3 months corrected age
Maternal side effects | Up to 3 months corrected age

OTHER OUTCOMES:
Costs | Up to 3 months corrected age

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam University Medical Centres, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Klumper J, Breebaart W, Roos C, Naaktgeboren CA, van der Post J, Bosmans J, van Kaam A, Schuit E, Mol BW, Baalman J, McAuliffe F, Thornton J, Kok M, Oudijk MA. Study protocol for a randomised trial for atosiban versus placebo in threatened preterm birth: the APOSTEL 8 study. BMJ Open. 2019 Nov 26;9(11):e029101. doi: 10.1136/bmjopen-2019-029101. PMID 31772083
- See also: Related Info — https://zorgevaluatienederland.nl/evaluations/apostel8